CLINICAL TRIAL: NCT04562324
Title: Efficacy of Electroencephalography (EEG) Neurofeedback (NF) of Motor Sensory Cortex as an Add-on Treatment for Drug-naïve Anxiety Disorder: A Randomized, Double-blind, Sham-controlled Trial
Brief Title: Efficacy of Electroencephalography (EEG) Neurofeedback (NF) for the Treatment of Anxiety Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NF-2020-TJAH
Record Dates: First submitted 2020-09-19; First posted 2020-09-24 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Anxiety Disorder; Healthy
MeSH Terms: conditions — Anxiety Disorders | interventions — Selective Serotonin Reuptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors; Benzodiazepines; Antidepressive Agents, Tricyclic; Antipsychotic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: (Experimental): NF group participants receive 24 min NF sessions over the Motor sensory Cortex, 2-3 days per week, for 2 weeks combine a selective serotonin reuptake inhibitor (SSRI) or a serotonin or norepinephrine reuptake inhibitors (SNRI) or benzodiazepines or tricyclic antidepressants or other antidepressants or antipsychotics or other sedative-hypnotics
  Interventions: Drug: SSRI or SNRI or benzodiazepines or tricyclic antidepressants or other antidepressants or antipsychotics or other sedative-hypnotics; Device: Neurofeedback system
- Healthy Experimental: (Experimental): Participants receive 24 min NF sessions over the Motor sensory Cortex, 2-3 days per week, for 2 weeks
  Interventions: Device: Neurofeedback system
- Healthy Sham Comparator (Sham Comparator): Sham group participants receive 24 min NF sessions with pseudo-random numbers, 2-3 days per week, for 2 weeks
  Interventions: Device: Neurofeedback system
- Sham Comparator (Sham Comparator): Sham Comparator: Sham group participants receive 24 min NF sessions with pseudo-random numbers, 2-3 days per week, for 2 weeks combine a selective serotonin reuptake inhibitor (SSRI) or a serotonin and norepinephrine reuptake inhibitors (SNRI), benzodiazepines, tricyclic antidepressants, other antidepressants, antipsychotics, other sedative-hypnotics
  Interventions: Drug: SSRI or SNRI or benzodiazepines or tricyclic antidepressants or other antidepressants or antipsychotics or other sedative-hypnotics; Device: Neurofeedback system

INTERVENTIONS:
Drug: SSRI or SNRI or benzodiazepines or tricyclic antidepressants or other antidepressants or antipsychotics or other sedative-hypnotics — Medications to relieve anxiety
  Arms: Experimental:; Sham Comparator
Device: Neurofeedback system — EEG-neurofeedback is an operant conditioning procedure in which people learn to improve the brain's functional activity and used as a way to effect long-term change in abnormal brain activity thus alter corresponding cognitive function. In addition, its potential to be used to elucidate the mechanisms underlying psychopathology by evaluating the subjective effect of the modulation of specific brain areas has become apparent. Participants receive 24 min NF sessions over the Motor sensory Cortex, 2-3 days per week, for 2 weeks

SUMMARY:
The aim of this study is to assess the efficacy of electroencephalography (EEG) neurofeedback (NF) as an Add-on Treatment for the Anxiety disorder. Meanwhile, evaluate the effect of EEG-NF on cognitive function of Anxiety patients. Furthermore, the investigators will examine the changes in cortisol, gut microbiome and some biomarkers. The hypothesis of this study is that EEG-NF alleviate the anxiety symptoms and improve the cognitive function of Anxiety disorder patients with regulating attention response.

DETAILED DESCRIPTION:
This is a randomized, double-blind, sham-controlled study using electroencephalography (EEG) neurofeedback (NF) for 2-week treatment. Participants were randomly assigned 1:1 to NF group or sham-control group. The NF group performed six NF sessions every other day in about two weeks. The feedback value of the NF group was about SMR band, while in the control group was pseudo-random numbers. Apart from studying the effects of EEG-NF on severity of anxiety and cognitive function, the secondary outcomes are to examine biomarkers related to inflammatory activity. Scale assessments are performed before the initiation of treatment, week 1, week 2. The Digit Span test, Go/No-Go task Collection of blood, excrement and saliva takes place at two time points, at the baseline, week 2.

ELIGIBILITY:
Inclusion Criteria:

* a current episode of Anxiety diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* age between 18 and 50 years
* a total score of HAMD ≥14 GAD-7≥ 5
* Participants are compliant with treatment according to the judgement of the treating clinician.
* Participant or guardian has to sign informed consent. The patients' guardians will sign the informed consent on behalf of the participants when the capacity of participants to consent is compromised.

Exclusion Criteria:

* History of alcohol or drug abuse;
* Severe somatic diseases including conditions such as kidney and liver failure, uncontrolled hypertension, cardiovascular, cerebrovascular and pulmonary disease, thyroid disease, diabetes, epilepsy and asthma.
* Use of anti-inflammatory medication for longer than 7 days in the last two months preceding the trial
* Use of immunosuppressive medication such as oral steroid hormones Women in pregnancy or lactation period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
The change of scores in Hamilton Anxiety Rating Scale (HAMD) from baseline to week 2. | baseline, Week 1, week 2
  The main objective is to explore whether NF add on medicine will improve the anxiety symptoms after 2 weeks of treatment, and investigators assess the scale at baseline and week 1, 2. Hamilton Anxiety Rating Scale (HAMD) items was used to evaluate the severity of symptoms of anxiety. A total score of more than 29 may indicate severe anxiety symptoms; A score above 14 may be mild to moderate anxiety; If the score is less than 7, the patient has no symptoms of anxiety. The higher the total score of the scale, the more severe the anxiety symptoms.
The change of scores in GAD-7 from baseline to week 2. | baseline, Week 1, week 2
  The main objective is to explore whether NF add on medicine will improve the anxiety symptoms after 2 weeks of treatment, and investigators assess the scale at baseline and week 1, 2. GAD-7 items were used to evaluate the severity of symptoms of anxiety. A total score of more than 15 may indicate severe anxiety symptoms; A score above 5 may be mild to moderate anxiety; If the score is less than 4, the patient has no symptoms of anxiety. The higher the total score of the scale, the more severe the anxiety symptoms.

SECONDARY OUTCOMES:
The change of scores in the State-Trait Anxiety Inventory (STAI) from baseline to week 2. | baseline, Week 1, week 2
  The main objective is to explore whether NF add on medicine will improve the anxiety symptoms after 2 weeks of treatment, and investigators assess the scale at baseline and week 1, 2. State-Trait Anxiety Inventory (STAI) items was used to evaluate the severity of symptoms of anxiety. The total score of STAI ranged from 20 to 80. The higher the score, the worse the severity of symptoms of anxiety.
The change of scores in Pittsburgh Sleep Quality Index (PSQI) from baseline to week 2. | baseline, Week 1, week2
  The aim is to investigate whether NF training in addition to regular treatment with medicine will improve the sleep quality as measured with Pittsburgh Sleep Quality Index (PSQI) after 2 weeks of treatment compared to sham-group, and investigators assess the scale at baseline, week1and week 2. PSQI was used to evaluate the sleep quality of the subjects in the latest month. The total score of PSQI ranged from 0 to 21. The higher the score, the worse the sleep quality.
The change of scores in Insomnia Severity Index (ISI) from baseline to week 2. | baseline, Week 1, week 2
  The aim is to investigate whether NF training in addition to regular treatment with medicine will improve the sleep quality as measured with Insomnia Severity Index (ISI) after 2 weeks of treatment compared to sham-group, and investigators assess the scale at baseline, week1and week 2. The ISI scale was used to evaluate the severity of insomnia. The higher the score, the more severe the insomnia
The change of scores in Mindful Attention Awareness Scale, MAAS) from baseline to week 2. | baseline, Week 1, week 2
  The aim is to investigate whether NF training in addition to regular treatment with medicine will improve the level of mental resilience, attention and consciousness as measured with Mindful Attention Awareness Scale, MAAS) after 2 weeks of treatment compared to sham-group, and investigators assess the scale at baseline, week1and week 2. The MAAS scale evaluates assess the level of mental resilience. The higher the score, the higher the participant's level of mindfulness.
The changes of levels of biomarkers in peripheral blood from baseline to week 2 | baseline, week 2
  The aim is to investigate the change of cortisol level of saliva and intestinal flora as active stimuli in addition to regular treatment with medicine after 2 weeks of treatment compared to sham group, and investigators collect the specimens at baseline and week 2.
  Saliva collection tube to collect saliva, collect naturally discharged saliva in a clean test tube (at least 2ml). Saliva was centrifuged under 1500rpm for 15 minutes and the filtrate was cryopreserved at-80 C. the saliva was analyzed by ELISA kit.
  Fecal collection: a) intercept the middle part of the sample with a sterile toothpick or fecal sampler (the surface of feces contains exfoliated cells of intestinal mucosa; the outside is easy to be contaminated, and some bacterial DNA begins to degrade after contact with air), take about the size of peanuts and put them into aseptic 2.0mL centrifuge tubes, 3-5 tubes for each sample are taken for backup#and then put into-80°C cryopreservation after sub-packaging.
Adverse events from baseline to week 2 | week 1, week 2
  2 The aim is to evaluate the adverse effects during the treatment.
The change of reaction time in Go/No-Go task from baseline to week 2. | baseline, week 2
  The aim is to investigate whether NF training in addition to regular treatment with medicine will improve attention as measured with Go/No-Go task after 2 weeks of treatment compared to sham-group, and investigators assess the scale at baseline and week 2. The Go/No-Go task scale evaluates assess the level of attention. The shorter the reaction time, the higher the level of attention.
The accuracy in the Digit Span test (DSP) from baseline to week 2. | baseline, week 2
  The aim is to investigate whether NF training in addition to regular treatment with medicine will improve short-term memory and working memory as measured with the Digit Span test (DSP) after 2 weeks of treatment compared to sham-group, and investigators assess the scale at baseline and week 2. The Digit Span test (DSP) scale evaluates assess short-term memory and working memory. The higher the accuracy, the better the level of memory.
The change of scores in Self-Rating Anxiety Scale (SAS) from baseline to week 2. | baseline, week 2
  The main objective is to explore whether NF will improve the anxiety symptoms after 2 weeks of treatment, and investigators assess the scale at baseline and week 2. Self-Rating Anxiety Scale (SAS)items was used to evaluate the severity of symptoms of anxiety. A total score of more than 56 may indicate severe anxiety symptoms; A score above 40 may be mild to moderate anxiety; If the score is less than 20, the patient has no symptoms of anxiety. The higher the total score of the scale, the more severe the anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided